CLINICAL TRIAL: NCT04042844
Title: A Phase 2, Double-Blind, Controlled, Randomized Study to Evaluate the Safety and Preliminary Efficacy of a Single Dose Intradiscal Injection of BRTX-100 for Patients With Chronic Lumbar Disc Disease (cLDD)
Brief Title: A Single Dose of BRTX 100 for Patients With Chronic Lumbar Disc Disease (cLDD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioRestorative Therapies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLDD-001
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Disc Disease
MeSH Terms: conditions — Intervertebral disc disease | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized (2:1) to receive either intradiscal BRTX-100 or control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment- BRTX-100 (Experimental): BRTX-100 consists of a population of hypoxic-cultured bone marrow mononuclear cells highly enriched in mesenchymal stem cells from autologous bone marrow with autologous platelet lysate.
  Interventions: Biological: BRTX-100
- Sham (Sham Comparator): Isotonic saline will be used as a control (sham) in this study. Drug: saline (0.9% sodium chloride).
  Please note this will be a sham procedure. This isotonic saline will not be injected intradiscally.
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: BRTX-100 — Hypoxic cultured mesenchymal stem cells (MSCs) from autologous bone marrow with autologous platelet lysate.
  Arms: Active Treatment- BRTX-100
Drug: Saline — Sodium Chloride (0.9%) intravenous infusion preparation is a sterile and non-pyrogenic solution
  Arms: Sham

SUMMARY:
This is a double-blind, controlled, randomized study with blinded assessments using a single dose. Subjects that have a current diagnosis of chronic lumbar disc disease and meet eligibility criteria will be enrolled. Chronic lumbar disc disease is defined as back and/or radicular pain with degeneration of the disc confirmed by patient history, physical examination, and radiographic measures such as computed tomography (CT), magnetic resonance imaging (MRI), plain film, myelography, discography, or other acceptable means.

DETAILED DESCRIPTION:
This is a double-blind, controlled, randomized study with blinded assessments using a single dose. Subjects that have a current diagnosis of chronic lumbar disc disease and meet eligibility criteria will be enrolled. Chronic lumbar disc disease is defined as back and/or radicular pain with degeneration of the disc confirmed by patient history, physical examination, and radiographic measures such as computed tomography (CT), magnetic resonance imaging (MRI), plain film, myelography, discography, or other acceptable means.

Subjects randomized to active treatment will undergo bone marrow harvest for processing into BRTX- 100 for intradiscal injection. Subjects randomized to control will also undergo a bone marrow and blood harvest but only undergo a sham intradiscal injection procedure. Subjects will return to the study site for a visit at Week 2, Week 12, Week 26, Week 52 and Week 104/Early Termination.

The trial will have a Safety Run-In component that will insert a 3+3 design for the initial subjects dosed with BRTX-100 at 40 × 10^6 cells. Specifically, the randomization scheme will be briefly shifted from the overall trial 2:1 randomization to an initial 3:1 allotment of intradiscal BRTX-100 versus control.

As such, four subjects will initially be randomized and administered their agents. There will be a 14-day safety follow-up period that must elapse between dosing of each of the first four (4) subjects. Dosing of each subsequent subject in the Safety Run-In component cannot occur until the independent Medical Monitor (MM) reviews the previously dosed subject's blinded data, including but not limited to physical examination findings, laboratory values and reported adverse events (AEs) and serious adverse events (SAEs), at the completion of the 14-day visit and documents the findings. If no potential dose-limiting toxicity (DLT) is noted by the MM, the MM will approve the dosing of the next subject. If a potential DLT is noted by the MM, the MM will request that an ad hoc Data Safety Monitoring Board (DSMB) review of unblinded data occur per DSMB Charter before the next subject is dosed.

ELIGIBILITY:
Subject Inclusion Criteria:

A subject is eligible for inclusion if all the following criteria are met:

1. A high index of suspicion for discogenic pain, (i.e., painful degenerative disc(s) with or without protrusions less than or equal to 5 mm)

   1. Chronic Lower Back Pain for at least 6 months
   2. Pain commonly provoked by prolonged sitting, forward bending, lifting, twisting, coughing, sneezing, or Valsalva maneuvers
   3. Failure of at least 6 months of conservative back pain care (can include any or all of the following: rest, anti-inflammatory medication, analgesics, narcotics, epidural injections or selective nerve root injections at the target level, facet joint injections, muscle relaxers, massage, acupuncture, chiropractic care)
   4. Failure of supervised therapy (such as physical therapy)
   5. Screening of ≥ 40 mm and ≤ 80 mm on low back pain visual analog scales (VAS) (average pain in the last week)
   6. Screening Oswestry Disability Index (ODI) score ≥ 30 and < 90 on a 100-point scale
   7. No localized and significant pain below beltline (i.e., potential sacroiliac joint pain) without lumbar pain component
   8. Thigh or Leg pain, if present, is non prevailing and of nonradicular origin, i.e., not due to stimulation of nerve roots or dorsal root ganglion of a spinal nerve by compressive forces
   9. Diagnostic medial branch block or facet joint injection (bilateral unless the symptoms are purely unilateral in nature) in the last 12 months prior to the informed consent date indicates no prevailing facet joint involvement
2. Has degenerative disc disease (DDD) as defined by the following:

   1. Changes from normal disc morphology of the affected disc as defined by radiographic evaluation
   2. Modified Pfirrmann score of 2 to 7 on MRI, may contain a contained protrusion and/or annular tear on MRI
   3. Modified Pfirrmann score of 1 must contain a contained protrusion and/or annular tear on MRI
   4. Modic Grade I or II changes or no change on MRI
   5. Maintained intervertebral disc heights of at least 50% on MRI.
   6. Discography, if not performed within the last 6 months prior to informed consent date, has to be performed if more than one degenerative disc is identified by MRI, and the symptomatic disc cannot be otherwise reasonably determined
   7. If more than one degenerative disc is identified by MRI, no disc shall demonstrate greater degenerative change than the symptomatic disc or contain a protrusion greater than 5mm
3. Aged ≥18 years of age at the time of consent
4. Willing and able to provide written informed consent
5. No evidence of contraindications to the procedure such as pregnancy, active infection, bleeding disorder, or metastatic cancer

Subject Exclusion Criteria:

A subject is not eligible to participate if any of the following criteria are met:

1. Spinal Deformity (Scoliosis greater than or equal to 20 degrees, spondylolysis, clinically or radiographically significant retrolisthesis or spondylolisthesis) detected on MRI or plain film radiographic assessment
2. Disc extrusions, sequestered fragments, facet cysts, or greater than moderate spinal stenosis on MRI.
3. Presence of a Grade V annular fissure observed within the index disc level during discography in a subject for whom provocation discography has been performed
4. Intervertebral disc with radiographic evidence of Modified Pfirrmann Grade 8 or greater
5. Any bleeding disorder, intrinsic or extrinsic
6. Required anticoagulation (with either antiplatelet agents or antithrombotics) that cannot be interrupted for harvest and injection procedures
7. Platelet count less than or equal to 100,000
8. International Normalized Ratio (INR) greater than or equal to 1.5
9. Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI greater than or equal to 40)
10. Clinically relevant instability on flexion-extension as determined by the investigator by overlaying films (flexion & extension films)
11. Has undergone any previous lumbosacral spine surgery (e.g. discectomy, laminectomy, foraminotomy, fusion, intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation.), ablation of lumbar basiverterbral nerve or therapeutic percutaneous disc intervention
12. Have any acute or chronic lumbosacral spine fracture
13. Have a history of lumbosacral epidural steroid injections within 1 month prior to informed consent date.
14. Planned/expected use of systemic nonsteroidal anti-inflammatory drugs (NSAIDs) within 72 hours prior to study treatment.
15. Have a known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO)
16. Active significant non lumbosacral spinal orthopedic pain generators including, not limited to arthritic hip and/or knee, cervical disc disease
17. More widespread and ill-defined myofascial pain
18. Have had treatment with any cellular or biological investigational therapy or device within 6 months of informed consent date and/or plans to participate in any other autologous or allogeneic stem cell/progenitor cell therapy trial during the 2 year follow-up period
19. Have been a recipient of any lumbosacral intervertebral disc injection for therapeutic purposes
20. Are transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program
21. Apparent ongoing and poorly controlled psychological or somatic disease that may impact treatment outcomes
22. Social, familial, or geographical hindrances to compliance with the study protocol or the informed consent process
23. Known autoimmune disease with primary impact on the musculoskeletal and/or neurological systems (e.g., systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, myasthenia gravis, polymyositis/dermatomyositis, Guillain-Barre syndrome, autoimmune vasculitis)
24. Required chronic immunosuppression
25. Positive hepatitis C virus (HCV) antibody test
26. Positive human immunodeficiency virus (HIV) Antigen/Antibody (Ag/Ab) Combo test
27. Pregnant or lactating women
28. Women of childbearing potential not protected by a highly effective method of birth control.

    Highly effective methods of contraception [defined as those, alone or in combination, that result in a low (<1%) failure rate] include, but are not limited to, combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (either oral, intravaginal, transdermal or injectable), progestogen-only hormonal contraception associated with inhibition of ovulation (either oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence, or a double-barrier method (i.e., male condom combined with diaphragm with spermicide). The investigator is responsible for review of medical history, contraception history, menstrual history and recent sexual activity to decrease the risk of including a woman with an undetected early pregnancy. Additionally, the investigator is responsible for determining if, in the investigator's judgment, a woman's planned contraceptive method (including an assessment of her reliability for consistent use of this method) meets the protocol requirement of "highly effective."
29. Hematology and chemistry values including, but not limited to:

    1. Total bilirubin level 1.5 times institutional upper limit of normal (ULN)
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2 x ULN
    3. Absolute neutrophil count (ANC) < 1000/mm3
    4. Hemoglobin less than or equal to 10 g/dL
    5. Creatinine clearance use calculated clearance (Cockcroft-Gault equation) of less than or equal to 50 mL/min
    6. Other labs deemed clinically significant which, in the opinion of the investigator, might influence the subject's health or safety during the trial.
30. Have any other active medical conditions, medical or psychiatric illness which, in the opinion of the Investigator, would preclude adequate evaluation of the safety and efficacy of the study or put the participant at risk
31. Inability to comply with the requirements of the study protocol
32. Actively on workers compensation or no-fault case for this complaint or any other active case or litigation pertaining to their lumbosacral pain.
33. History of drug or alcohol abuse or documented history of noncompliance with controlled substances that, in the investigator's opinion, could interfere with adequate evaluation of the study drug's safety or efficacy or otherwise make the subject unsuitable for the study.
34. History of regular, long term, daily opioid drug use (greater than or equal to 30 MME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Measures | Baseline through Week 104 / Early Termination
  Report of adverse events (AEs), clinical review and questionnaires for pain, disability and quality of life at Baseline through Week 104/ Early Termination
  * Vital Signs
  * Physical Examination
  * Laboratory Evaluation (hematology and chemistry)
  * Clinical review of MRI changes from Baseline to Week 104 (MRI density measurements in T2 weighted images performed at Baseline, Week 52 and Week 104 with predetermined MRI rating scores)
Primary Efficacy Measures | Baseline through Week 52
  * VAS for Pain Assessment
  * ODI for Functional Assessment
  Primary Efficacy Endpoint:
  Clinical response, defined as at least a 30% decrease in pain as measured on the VAS scale and at least a 30% increase in function based on the ODI at Week 52 as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lipitz, MD, Study Chair — BioRestorative Therapies
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Source Healthcare, Santa Monica, California
  - Boomerang Healthcare, Walnut Creek, California
  - Denver Back Pain Specialists, LLC, Greenwood Village, Colorado
  - Cantor Spine Institute, Fort Lauderdale, Florida
  - Coastal Health, Jacksonville, Florida
  - Pain Relief Centers, St. Petersburg, Florida
  - Tampa Pain Relief Center, Tampa, Florida
  - Florida Pain Relief Center, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Northwell Health, New York, New York
  - The Center of Clinical Research, LLC, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Investigations LLC, Edmond, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Science Connections, Austin, Texas
  - NCP Center for Clinical Research and Innovation, Houston, Texas
  - Precision Spine Care, Tyler, Texas
  - Virginia iSpine Physicians, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No